CLINICAL TRIAL: NCT03836144
Title: Effect of Urine Alkalinazation on Urinary Inflammatory Markers Analyzed Using Mass Spectrometry in Patients With Cystinuria
Brief Title: Effect of Urine Alkalinazation on Urinary Inflammatory Markers in Patients With Cystinuria
Status: Completed | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Sponsor Name Pending (Industry)
Responsible Party: Principal Investigator, Marie Courbebaisse, Associate Professor, MD, PhD, European Georges Pompidou Hospital
Other Study IDs: EuropeanGPH
Record Dates: First submitted 2019-01-21; First posted 2019-02-11 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Cystinuria; Renal Lithiasis; Glomerulonephritis; Interstitial Nephritis
Keywords: Mass spectrometry; Cystinuria; Inflammation; Nephrolithiasis
MeSH Terms: conditions — Cystinuria; Nephrolithiasis; Glomerulonephritis; Nephritis, Interstitial; Inflammation | interventions — Potassium Citrate; Sodium Bicarbonate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cystinuria: 10 patients with cystinuria. Experimental. Urine collected before treatment initiation and 3 months after. Treatment: Usual alkalizing treatment using oral potassium citrate. The initial dosage will be 4 g/day divided into 3 to 4 oral daily doses. If the objective of urinary pH is not reached after the first two weeks of treatment, the dose will be increased by 2 grams (6 grams total). If the urinary pH remains below 7.5 after 2 weeks with 6 grams of potassium citrate per day, the alkalizing treatment will then be supplemented with oral sodium bicarbonate in the form of Vichy water or officinal preparation. This treatment is the usual treatment recommended for cystinuria .
  Interventions: Dietary Supplement: Potassium citrate
- Non cystinuria nephrolithiasis: 20 patients with a nephrolithiasis not due to cystinuria. Control group. Urine collected once to study biomarkers of inflammation No intervention.
- Inflammatory nephropathy: 10 patients with an inflammatory nephropathy of glomerular or tubulo interstitial origin (confirmed by renal biopsy).
  Control group. Urine collected once to study biomarkers of inflammation. No intervention.

INTERVENTIONS:
Dietary Supplement: Potassium citrate
  Other Names: Sodium bicarbonate
  Groups: Cystinuria

SUMMARY:
It has recently been described the presence of a urinary inflammatory signature in patients with cystinuria, the most common cause of renal lithiasis of genetical origin. These data are very innovative in this pathology but deserve further studies to establish the specificity of this inflammatory signature in patients with cystinuria compared to other nephropathies and other renal lithiasis diseases. Moreover, the effect of the usual treatment of cystinuria (namely urine alkalanization) on urinary inflammatory biomarkers deserves to be tested.

The objectives of the present study are: i) To study the urinary inflammatory profile by mass spectrometry (a very efficient tool to detect and identify proteins) in patients with cystinuria and in patients with lithiasis of other origin and in patients with inflammatory renal disease ; ii) To study the potential effect of urine alkalinazation with potassium citrate (usual treatment according to European recommendations) on the inflammatory signature of patients with cystinuria. To this aim, urine of non treated cystinuric patients will be collected before treatement initiation and 3 months after the start of the alkalizing treatment.

ELIGIBILITY:
Inclusion Criteria:

* age superior or equal to 18 years
* patient able to understand the information note and to sign the informed consent
* patient with an Health coverage
* no current urinary tract infection (assessed by a cytobacteriological examination of the urine)
* For the cystinuria group: patient with cystinuria not yet treated or for whom the alkalizing treatment or the cystein binding thiol agents have been discontinuated for at least 3 months AND with an estimated GFR (using the MDRD formula) greater than 60 ml/min/1.73m2.
* For the control groups: patient presenting either a renal lithiasis not due to cystinuria, or an inflammatory renal pathology confirmed by an anterior renal biopsy (glomerulonephritis or interstitial nephritis) AND with an estimated GFR (using the MDRD formula) greater than 30 ml/ min/1.73m2.

Exclusion Criteria:

* Cystinuric patient already treated (whatever the treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cystinuria, as well as patients with renal lithiasis not due to cystinuria and patients with an inflammatory renal pathology will be selected by the investigators of the study during their usual medical consultation.
  At that time, patients will be given the information note and will be asked to sign the written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline urine inflammatory profile after 3 months of alkalizing treatment using mass spectrometry in patients with cystinuria. | at inclusion and after three months of the usual alkalizing treatment for the patients with cystinuria
  Study of urine inflammatory biomarkers profile using mass spectrometry to determine if the alkalizing treatment is susceptible to modify the urine inflammatory profile. Proteases inhibitors will be added to the urine sample immediately after urination. Urine will then be frozen at -80°C until mass spectrometry analysis. Mass spectrometry will determine the differential expression of all the proteins present the urine sample. For the purpose of the present study, the investigators will focus on the expression of inflammatory biomarkers among them MMP9 (matrix metallopeptidase), Myeloperoxydase, Proteinase 3, Neutrophil Elastase, Cathepsine G, LSP1 (lymphocyte specific protein), Fibrinogen beta and gamma chains. The aim of mass spectrometry is to detect the presence of proteins in the urine sample and to assess the differential levels of expression of the detected proteins but not to precisely measure the urine concentration of the detected proteins.

SECONDARY OUTCOMES:
Assessment of urine inflammatory profile in controls groups using mass spectrometry. | at inclusion for patients with a nephrolithiasis not due to cystinuria and in patients an inflammatory nephropathy of glomerular or tubulo interstitial origin
  Study of urine inflammatory biomarkers with mass spectrometry in control groups to determine if the urine inflammatory profile is specific to cystinuria. Proteases inhibitors will be added to the urine sample immediately after urination. Urine will then be frozen at -80°C until analysis. Mass spectrometry will determine the differential expression of all the proteins present the urine sample. For the purpose of the present study, the investigators will focus on the expression of inflammatory biomarkers. The aim of mass spectrometry is to detect the presence of proteins in the urine sample and to assess the differential levels of expression of the detected proteins but not to precisely measure the urine concentration of these proteins. Moreover, urine analysis by mass spectrometry will detect all urinary proteins and the investgators do exclude to find unexpected proteins. For those reasons, urine analysis by mass spectrometry is a unique outcome.
Study of crystalluria (presence of crystals in urine) to assess nephrolithiasis activity. | at inclusion for these two groups and after three months of the usual alkalizing treatment for the patients with cystinuria
  Assessment of the presence of crystals in the second morning urine sample in patients with cystinuria and in patients with a nephrolithiasis not due to cystinuria, to assess nephrolithiasis activity.

OTHER OUTCOMES:
Presence of stones in the renal cavities or in the urinary tract using ultrasonograhy. | at inclusion for these two groups and after three months of the usual alkalizing treatment for the patients with cystinuria
  assessment of the presence of urinary stones using ultrasonogrpahy in patients with cystinuria and in patients with a nephrolithiasis not due to cystinuria.
Blood CRP concentrations to assess systemic inflammation | at inclusion for all groups and and after three months of the usual alkalizing treatment for the patients with cystinuria
  Blood CRP concentration (mg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurpean Georges Pompidou Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bourderioux M, Nguyen-Khoa T, Chhuon C, Jeanson L, Tondelier D, Walczak M, Ollero M, Bekri S, Knebelmann B, Escudier E, Escudier B, Edelman A, Guerrera IC. A new workflow for proteomic analysis of urinary exosomes and assessment in cystinuria patients. J Proteome Res. 2015 Jan 2;14(1):567-77. doi: 10.1021/pr501003q. Epub 2014 Nov 12. PMID 25365230
- [Result] Prot-Bertoye C, Lebbah S, Daudon M, Tostivint I, Bataille P, Bridoux F, Brignon P, Choquenet C, Cochat P, Combe C, Conort P, Decramer S, Dore B, Dussol B, Essig M, Gaunez N, Joly D, Le Toquin-Bernard S, Mejean A, Meria P, Morin D, N'Guyen HV, Noel C, Normand M, Pietak M, Ronco P, Saussine C, Tsimaratos M, Friedlander G, Traxer O, Knebelmann B, Courbebaisse M; French Cystinuria Group. CKD and Its Risk Factors among Patients with Cystinuria. Clin J Am Soc Nephrol. 2015 May 7;10(5):842-51. doi: 10.2215/CJN.06680714. Epub 2015 Feb 25. PMID 25717071